CLINICAL TRIAL: NCT02448069
Title: ARTSS-IA: A Pilot, Phase IIa, Safety and Feasibility Study of ARgatroban in Combination With Recombinant Tissue Plasminogen Activator Stroke Study - Intra-Arterial
Brief Title: Safety and Feasibility of Argatroban, Tissue Plasminogen Activator and Intra-arterial Therapy in Stroke
Acronym: ARTSS-IA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Andrew D. Barreto, MD, MD, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0327
Record Dates: First submitted 2015-05-11; First posted 2015-05-19 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Stroke; Cerebral Ischemia
MeSH Terms: conditions — Stroke; Brain Ischemia | interventions — argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Argatroban treatment (Experimental): Intravenous Argatroban delivered at 100mcg/kg bolus, then 12-hour infusion initiated at 3mcg/kg/min.
  Interventions: Drug: Argatroban

INTERVENTIONS:
Drug: Argatroban — All patients will receive a 3.0 mcg/kg/min continuous infusion of Argatroban, preceded by a 100 mcg/kg bolus. Infusion will be titrated to achieve an aPTT of 2.25 times baseline (not to exceed 10 mcg/kg/min) for a maximum of 12 hours.

SUMMARY:
Background:

Our prior work with combination argatroban + recombinant tissue plasminogen activator (rt-PA) (ARTSS-1: Phase IIa low-dose safety study; n=65 and ARTSS-2: Phase IIb randomized low and high-dose study; n=90), demonstrated safety of the two drugs when delivered concomitantly and recanalization rates were greater than with historical controls. Further, interim analysis of neurological outcomes at 75 patients of the randomized Phase IIb trial, demonstrated a signal of efficacy when compared to control (rt-PA alone) patients. However, rt-PA fails to reperfuse brain in most patients with large thrombi, prompting several recent randomized clinical trials which have demonstrated that intra-arterial therapy (IA) following rt-PA substantially improves outcome in patients with distal carotid or proximal middle cerebral artery occlusions. As a result, rt-PA + IA has become the new standard-of-care for many patients with large arterial occlusions such as those treated in ARTSS-1 and 2. Therefore, this study is necessary to explore the feasibility and safety of adding Argatroban in acute ischemic stroke patients who also receive rt-PA followed by IA.

Primary Objective:

To demonstrate the feasibility and safety of treating stroke patients with Argatroban who undergo usual thrombolysis care (intravenous rt-PA followed by IA).

Secondary Objectives:

1. Assess rates of ultra-early recanalization at commencement of IA;
2. Assess the completeness and pattern of reperfusion as obtained by IA; 3) Assess clinical outcome

DETAILED DESCRIPTION:
Design:

Prospective, single-arm, open-label, feasibility and safety Phase IIa study.

Study Population:

10 total ischemic stroke patients all treated with rt-PA (0-3 hour or 0-4.5 hour according to each site's local standard) and IA; age of 18 years or older; proximal (intracranial) artery occlusion as imaged by CT-angiogram (CTA).

Treatment:

All patients will receive standard-of-care intravenous rt-PA (0.9 mg/kg; maximum 90 mg) and IA. Before the end of the 1 hour rt-PA infusion, a 3.0 mcg/kg/min continuous infusion of Argatroban, preceded by a 100 mcg/kg bolus will be administered over 3-5 minutes. Infusion will be titrated to achieve an aPTT of 2.25 times baseline (not to exceed 10 mcg/kg/min) for a maximum of 12 hours.

Assessments:

1. Baseline: History and physical exam, vital signs, CBC, liver function tests, PT/INR, PTT, non-contrast head CT, CT-Angiogram, NIHSS, mRS, concomitant medications.

   Laboratory results must be reported before study drug administration.
2. 0-24 hours: Vital signs, aPTT (scheduled 2, 6, 12 hours), NIHSS (24-hours), conventional angiography as part of usual care intra-arterial therapy. Repeat parenchymal brain imaging (non-contrast head CT or MRI) at 24 hours from rt-PA bolus. Laboratory testing work (same as baseline).
3. Day 7/Discharge (whichever occurs first): Vital signs, mRS, NIHSS
4. Day 90: mRS (obtained by certified rater).

ELIGIBILITY:
Inclusion Criteria:

* Disabling Ischemic stroke symptoms with onset < 3 hours treated with IV rt-PA by local standards*.

  * or </= 4.5 hours according to local standard of care. Symptoms must be distinguished from another ischemic event such as syncope, seizure, migraine, subarachnoid hemorrhage and hypoglycemia. If the patient reports awakening with the event, the time of onset should be considered as the last time the patient (or a witness to the patient's condition) considered herself/himself normal.
* Patients should meet local, institutional criteria to undergo emergent Endovascular Therapy (Intra-Arterial) to include:

  1. IAT must be able to begin before 6-hours of stroke onset or last seen well.
  2. CT-Angiogram confirmation of intra-arterial occlusion in any of the following locations: terminal ICA, MCA (M1 or M2 territories), PCA, distal vertebral or basilar artery.
  3. ASPECTS score on non-contrast head CT must be >/= 6.
  4. IAT must be able to begin within 90 minutes of qualifying CT scan.
* Age >/= 18.
* Females of childbearing potential must have a negative pregnancy test prior to the administration of trial medication.
* Signed (written) informed consent by the patient or the patient's legal representative and/or guardian.

Exclusion Criteria:

* Evidence of intracranial hemorrhage (ICH) on baseline CT scan or diagnosis of a non-vascular cause of neurologic deficit.
* NIHSS Level of Consciousness score (1a) >/= 2.
* Pre-existing disability with mRS > 2.
* Any evidence of clinically significant bleeding, or known coagulopathy.
* INR >1.5.
* Patients with an elevated aPTT greater than the upper limit of normal (test can be repeated if investigator suspects a falsely elevated value such as when the collection tube is not completely filled).
* Patients currently, or within the previous 24 hours, on an oral direct thrombin inhibitor (i.e., dabigatran), a factor 10a inhibitor (i.e., rivaroxaban, apixaban), or any other long-acting anticoagulant.
* Heparin flush required for an IV line. Line flushes with saline only.
* Any history of intra-cranial hemorrhage, known ateriovenous-malformation or unsecured cerebral aneurysms.
* Significant bleeding episode [e.g. gastrointestinal (GI) or urinary tract] within the 3 weeks before study enrollment.
* Major surgery or serious trauma in last 2 weeks. - Patients who have had an arterial puncture at a non-compressible site, biopsy of parenchymal organ, or lumbar puncture within the last 2 weeks.
* Previous stroke, myocardial infarction (MI), post myocardial infarction pericarditis, intracranial surgery, or significant head trauma within 3 months.
* Uncontrolled hypertension (SBP > 185 mmHg or DBP >110 mmHg) that does not respond to intravenous anti-hypertensive agents.
* Surgical intervention (any reason) anticipated within the next 48 hours.
* Known history of clinically significant hepatic dysfunction or liver disease - including a current history of alcohol abuse.
* Abnormal blood glucose <50 mg/dL (2.7 mmol/L).
* History of primary or metastatic brain tumor.
* Current platelet count < 100,000/mm3.
* Life expectancy < 3 months.
* Patients who, in the judgment of the investigator, needs to be on concomitant (i.e., during the Argatroban infusion) anticoagulants other than Argatroban, including any form of heparin, UFH, LMWH, defibrinogenating agent, dextran, other direct thrombin inhibitors or thrombolytic agents, GPIIb/IIIa inhibitor or warfarin. [*Caveat: However, if in the judgment of the investigator a patient needs to be anticoagulated, but this can be deferred for 48 hours, then they could be included.]
* Currently participating or has participated in any investigational drug or device study within 30 days before the first dose of study medication.
* Known hypersensitivity to Argatroban or its agents.
* Additional exclusion criteria if patient presents between 3-4.5 hours:

  1. Age >80
  2. Currently taking oral anticoagulants (regardless of INR)
  3. A history of stroke and diabetes.
  4. NIHSS > 25.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the incidence (absolute number) of symptomatic intracranial hemorrhage (sICH) | 12-36 hours after rt-PA bolus.
  defined as:
  1. Any evidence of bleeding on brain imaging that is associated with clinically significant neurological worsening (Greater or equals 4 NIH stroke scale points) and
  2. Parenchymal Hemorrhage 2 (PH-2); evidence of confluent hemorrhage on brain imaging that occupies > 30% of the volume of the infarct and produces significant mass effect.

SECONDARY OUTCOMES:
Feasibility of combining Argatroban with usual care as measured by success of starting the study medication bolus before the end of rt-PA infusion. 1. CT to tPA time, 2. CT to groin-puncture compared to institutional stroke-center database | 0-12 hours after stroke onset or hospital presentation.
Safety as measured by the incidence (absolute number of cases) of: 1. Groin or retroperitoneal hematoma 2. Major systemic hemorrhage requiring transfusion 3. Arterial perforation or dissection | 0-48 hours after enrollment.
Rates and completeness of arterial reperfusion as measured by cerebral angiography. Assessed at time of diagnostic (first intracranial injection unilateral to the occlusive lesion) and at the termination of study procedure. | At the end of Intra-Arterial therapy procedure (usually <12 hours from enrollment)
A NIH Stroke Scale (NIHSS) assessment will be performed at baseline and repeated at 24 hours, 48 hours and Day 7/discharge (whichever comes first). | 24, 48 hours, and Day 7 after rt-PA treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Barreto, MD, MS, Principal Investigator — UT HEalth Sicience Center, Houston Medical School, Department of Neurology, Stroke Team
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States